CLINICAL TRIAL: NCT04957550
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Phase 3 Clinical Study to Evaluate the Efficacy and Safety of SHR0302 in Active Psoriatic Arthritis Subjects
Brief Title: To Evaluate the Efficacy and Safety of SHR0302 Tablet in Subjects of Active Psoriatic Arthritis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0302-303
Record Dates: First submitted 2021-07-05; First posted 2021-07-12 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: SHR0302 tablets compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental): SHR0302 tablets dose 1+ Placebo dose 2
  Interventions: Drug: SHR0302 tablets、Placebo
- Treatment group B (Experimental): SHR0302 tablets dose 2+ Placebo dose 1
  Interventions: Drug: SHR0302 tablets、Placebo
- Treatment group C (Placebo Comparator): Placebo dose1 + placebo dose 2
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR0302 tablets、Placebo — SHR0302 tablets dose 1 for 48 weeks
  Arms: Treatment group A
Drug: SHR0302 tablets、Placebo — SHR0302 tablets dose 2 for 48 weeks
  Arms: Treatment group B
Drug: Placebo — SHR0302 tablets blank preparation for 24 weeks then SHR0302 tablets dose 1/dose 2 for 24 weeks
  Arms: Treatment group C

SUMMARY:
This study is a phase 3 study,to evaluate the efficacy and safety of different doses of JAK1 inhibitor SHR0302 in subjects with active psoriatic arthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Provide signed informed consent；
2. Diagnosis of PsA fulfillment of the Classification Criteria for PsA (CASPAR) criteria with symptom onset at least 6 months prior to the Screening Visit；
3. Active arthritis at screening/baseline as indicated by >/= 3 tender/painful and 3 swollen joints；
4. Diagnosis of active plaque psoriasis or documented history of plaque psoriasis.

Exclusion Criteria:

1. History of other autoimmune diseases; history of cancer or infection including tuberculosis and hepatitis; history of important cardiovascular events or thrombotic diseases；
2. Non-plaque forms of psoriasis (with exception of nail psoriasis)；
3. Previous treatment with cytotoxic drugs; JAK inhibitor or bDMARDs within 6 months of randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2024-11-13 (Estimated); Study Completion 2024-11-13 (Estimated)

PRIMARY OUTCOMES:
ACR20 response rate at week 24 | Week 24
  Percentage of Participants Meeting American College of Rheumatology Response Criteria Greater Than or Equal to (≥) 20% (ACR20) at week 24

SECONDARY OUTCOMES:
ACR20 response rate at week 48 | Week 48
  Percentage of Participants Meeting American College of Rheumatology Response Criteria Greater Than or Equal to (≥) 20% (ACR20) at week 48
ACR50/70 response rate at week 24 and week 48 | Week 24 and week48
  Percentage of Participants Meeting American College of Rheumatology Response Criteria Greater Than or Equal to (≥) 50%/70% (ACR50/70) at week 24 and week 48
Change from baseline in DAS28-CRP week 24 and week 48 | Week 24 and week 48
  Change from baseline in the disease activity score-CRP(DAS 28-CRP) at week 24 and week 48

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided